CLINICAL TRIAL: NCT05028517
Title: Efficacy Trial of the FMF Connect Mobile Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Research Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006555; U01AA026104 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Intervention Model Description: This study involves a three arm randomized controlled trial with equal allocation to the following conditions: (1) FMF Connect + coaching, (2) FMF Connect alone, and (3) waitlist control. Quantitative survey data will be collected at three timepoints: baseline (T1), 6-weeks (T2), and 12-weeks (T3).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMF Connect Intervention + Coaching (Experimental): Participants receive the FMF Connect mobile health app plus text-based coaching to support continued use of the app and individualized goal setting.
  Interventions: Other: FMF Connect; Other: Coaching
- FMF Connect Intervention (no coaching) (Experimental): Participants receive the FMF Connect mobile health app. They do not receive coaching.
  Interventions: Other: FMF Connect
- Waitlist comparison group (No Intervention): Participants receive the FMF Connect mobile health app at the conclusion of the study.

INTERVENTIONS:
Other: FMF Connect — The FMF Connect intervention includes cloud infrastructure and an innovative, multilayered mobile app. It incorporates tailored content for parents/caregivers of children (ages 3-12) with FASD or PAE. The app integrates five main components: 1) Dashboard; 2) Learning Modules; 3) Family Forum; 4) Library; and 5) Notebook. Weekly emails are also sent to support motivational engagement.
  Arms: FMF Connect Intervention (no coaching); FMF Connect Intervention + Coaching
Other: Coaching — A text-based coaching module is added to the FMF Connect app. Coaches support continued use of the app and individualized goal setting.
  Arms: FMF Connect Intervention + Coaching

SUMMARY:
The purpose of this study is to test a new smartphone "app" for parents/caregivers of children with fetal alcohol spectrum disorder (FASD). The app is called Families Moving Forward (FMF) Connect. The goal of the app is to provide parents/caregivers with useful information to help manage their children's condition and obtain peer support.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent or other primary caregiver (e.g., foster or adoptive parent, relative, legal guardian) of a child with FASD or prenatal alcohol exposure (PAE)
* The parent/caregiver must be at least 18 years old
* The child must between the ages of 3 and 12 years old
* The child has a diagnosis of FASD or has confirmed PAE
* The child has lived with the parent/caregiver for at least 4 months and is expected to remain in the home for at least 1 year
* The parent/caregiver lives in the United States
* The parent/caregiver has a smartphone or ipad with iOS operating system

Exclusion Criteria:

* The parent/caregiver is not fluent in English (the FMF Connect app and pre-post measures are currently only available in English)
* There is another parent/caregiver of the same child or living in the home that is already enrolled in the study (couples are excluded to prevent dependence in the data)
* The family has previously received or is currently receiving the therapist-led Families Moving Forward (FMF) Program - The caregiver participated in a prior trial of the FMF Connect app as part of earlier development phases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is deposited quarterly into the Collaborative Initiative on Fetal Alcohol Spectrum Disorders central repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be available once the data is collected and will be available indefinitely.
URL: http://www.cifasd.org/data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were asked to complete an eConsent and several screening questionnaires in REDCap. A total of 401 started the eConsent process. 272 were excluded for the following reasons: 37 did not meet inclusion criteria, 228 were incomplete, and 7 were duplicates.
Period: Overall Study
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Started | 43 | 43 | 43
Completed baseline surveys | 41 | 39 | 39
Completed 6-week follow-up surveys | 30 | 28 | 32
Completed (12-week Follow-up Surveys) | 30 | 23 | 30
Not Completed | 13 | 20 | 13
Not completed — Lost to Follow-up | 13 | 20 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 129 participants enrolled in the study and were allocated to the 3 arms. Demographic variables were provided at study enrollment. Data is available for demographics (age, sex, race, ethnicity, region) for 129 participants (43 per study arm). 10 participants did not complete baseline surveys, resulting in 119 participants with data for survey measures (Eyberg Child Behavior Inventory, Reasons for Children's Behavior, Parenting Sense of Competence, Family Needs Met, FASD Knowledge).
Groups:
- Total: Total of all reporting groups
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (7.0) | 43.1 (7.6) | 43.7 (7.6) | 44.00 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 40 | 124
  Male | 0 | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 41 | 43 | 40 | 124
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 00 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 40 | 41 | 39 | 120
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 43 | 129
Eyberg Child Behavior Inventory - Intensity Scale [Mean (Standard Deviation); unit: T-score] — The Eyberg Child Behavior Inventory measures the intensity of child behavior problems. Scores are presented as T-scores with a mean of 50 and a standard deviation of 10. A T-score of 60 or higher is considered clinically significant. Higher scores indicate more intense behavior problems. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in data available for FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  T-score
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 69.20 (8.86) | 69.51 (7.14) | 68.28 (9.01) | 69.00 (8.33)
Reasons for Children's Behavior Scale - Sensory Avoid [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Sensory Avoid scale measures attributions of behavior based on sensory avoidance. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in data available for FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 16.20 (5.32) | 19.18 (5.99) | 15.64 (6.06) | 16.99 (5.95)
Reasons for Children's Behavior Scale - Sensory Seek [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Sensory Seek scale measures attributions of behavior based on sensory seeking. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 23.15 (6.43) | 23.90 (4.98) | 22.56 (6.69) | 23.20 (6.06)
Reasons for Children's Behavior Scale - Task Willful [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Task Willful scale measures attributions of behavior based on willful task avoidance. It ranges from 3 to 18 with higher scores reflecting greater agreement with willful attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 10.51 (3.15) | 10.51 (2.89) | 10.05 (3.33) | 10.36 (3.11)
Reasons for Children's Behavior Scale - Task Ability [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Task Ability scale measures attributions of behavior based on ability to complete tasks. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 22.95 (4.61) | 23.67 (4.53) | 22.13 (4.26) | 23.57 (4.46)
Reasons for Children's Behavior Scale - Disruptive Behavior [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Disruptive Behavior scale measures attributions of behavior based on purposeful disruptive behavior. It ranges from 5 to 30 with higher scores reflecting greater agreement with willful attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 16.10 (6.24) | 15.36 (6.32) | 15.26 (7.37) | 15.56 (6.61)
Reasons for Children's Behavior Scale - Emotional Support [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Emotional Support scale measures attributions of behavior based on need for emotional support. It ranges from 4 to 24 with higher scores reflecting greater agreement with neurodevelopmental attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 19.68 (3.86) | 20.82 (3.04) | 20.90 (3.55) | 20.45 (3.52)
Reasons for Children's Behavior Scale - Dysregulated [Mean (Standard Deviation); unit: units on a scale] — The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Dysregulated Behavior scale measures attributions of behavior based on dysregulated behavior. It ranges from 3 to 18 with higher scores reflecting greater agreement with neurodevelopmental attributions. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 8.83 (3.87) | 9.56 (3.43) | 8.79 (3.57) | 9.06 (3.62)
Parenting Sense of Competence Scale - Efficacy [Mean (Standard Deviation); unit: units on a scale] — The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The efficacy sub-scale reported here measures how effective parents feel they are and includes 7 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 7 to 42 with higher scores indicating lower feelings of efficacy. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 26.78 (5.56) | 26.77 (5.18) | 25.23 (6.58) | 26.27 (5.79)
Parenting Sense of Competence Scale - Satisfaction [Mean (Standard Deviation); unit: units on a scale] — The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The satisfaction sub-scale reported here includes 9 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 9 to 54 with higher scores indicating higher satisfaction in the parenting role. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 34.12 (6.93) | 34.05 (7.85) | 33.41 (6.98) | 33.87 (7.20)
Family Needs Met Scale [Mean (Standard Deviation); unit: units on a scale] — The family needs questionnaire measures the degree to which family needs are met. The scale includes 18 items reflecting family needs that are rated on a scale from 0 to 4, with 0 being not applicable to 4 being met a great deal. The total score on this measure is created by summing across all items. Total score ranges from 0-72. Higher scores reflect more needs being met. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 39.93 (10.28) | 38.64 (10.77) | 38.44 (9.62) | 39.02 (10.17)
Knowledge and Advocacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Knowledge and Advocacy questionnaire assesses caregiver knowledge about FASD and advocacy and ranges from 0 to 28. Higher scores reflect greater knowledge. Population: A total of 129 participants were allocated to the 3 arms. A total of 10 did not complete baseline surveys, resulting in FMF Connect + Coaching = 41, FMF Connect (no coaching) = 39, and Waitlist = 39.
  units on a scale
    number analyzed (Participants) | 41 | 39 | 39 | 119
    (all) | 20.56 (2.59) | 20.97 (3.38) | 20.77 (3.65) | 20.76 (3.20)

OUTCOME MEASURES:

1. Primary Outcome: Eyberg Child Behavior Inventory - Intensity at Baseline and 12-week Follow-Up
Description: The Eyberg Child Behavior Inventory measures the intensity of child behavior problems. Scores are presented as T-scores with a mean of 50 and a standard deviation of 10. A T-score of 60 or higher is considered clinically significant. Higher scores indicate more intense behavior problems.
Time Frame: baseline to 12 weeks
Population: Data was analyzed from participants with complete data on the measure from both timepoints.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 30 | 23 | 30
T-score
  Baseline | 68.33 (1.65) | 69.13 (1.88) | 68.40 (1.65)
  12-week Follow-up | 64.47 (1.67) | 65.87 (1.90) | 66.03 (1.67)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; Mean comparisons of 3 separate groups using repeated measures ANOVA, including baseline and 12 week data. Participants with missing data were excluded. All participants were retained in their originally assigned group regardless of app usage; Test type: Superiority; p = .602, ANOVA; ANOVA Omnibus F test = 0.511
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; The FMF Connect + Coaching and FMF Connect groups were aggregated for analyses. Analyses were intent-to-treat, including all participants assigned to condition. Full information maximum likelihood (FMIL) was used for missing data in MPlus. Baseline and FMF Connect group status were entered into the regression model simultaneously. The dependent variable entered was the measure at the 12-week follow-up to determine treatment effects; Test type: Superiority; p = .33, Regression, Linear — False discovery rate (FDR) correction for multiple comparisons, p=.334; Cohen's d = -0.22, 95% CI 2-sided [-0.69 to 0.23]

2. Primary Outcome: Reasons for Children's Behavior - Sensory Avoid Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Sensory Avoid scale measures attributions of behavior based on sensory avoidance. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 15.54 (1.02) | 18.91 (1.17) | 16.57 (1.01)
  6-Week Follow-up | 15.87 (1.25) | 19.29 (1.45) | 18.25 (1.25)
  12-Week Follow-up | 15.43 (1.29) | 17.29 (1.49) | 17.57 (1.29)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; Mean comparisons of 3 separate groups using repeated measures ANOVA, including baseline, 6 week, and 12 week data. Participants with missing data were excluded. All participants were retained in their originally assigned group regardless of app usage; Test type: Superiority; p = .294, ANOVA; ANOVA Omnibus F test = 1.245
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; The FMF Connect + Coaching and FMF Connect groups were aggregated for analyses. Analyses were intent-to-treat, including all participants assigned to condition. Multiple imputation was used for missing data in SPSS. Analyses utilized linear mixed modeling for variables collected at the three timepoints; Test type: Superiority; p = .524, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.602; F(2) = .652

3. Primary Outcome: Reasons for Children's Behavior - Sensory Seek Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Sensory Seek scale measures attributions of behavior based on sensory seeking. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 23.79 (1.06) | 23.24 (1.23) | 23.29 (1.06)
  6-Week Follow-up | 23.36 (1.02) | 25.43 (1.17) | 24.39 (1.02)
  12-Week Follow-up | 22.61 (1.19) | 24.76 (1.37) | 23.14 (1.19)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .039, ANOVA; Anova Omnibus F test = 2.585
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; The FMF Connect + Coaching and FMF Connect groups were aggregated for analyses. Analyses were intent-to-treat, including all participants assigned to condition. Multiple imputation was used for missing data. Analyses utilized linear mixed modeling for variables collected at the three timepoints; Test type: Superiority; p = .548, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.893; F(2) = .606

4. Primary Outcome: Reasons for Children's Behavior - Task Willful Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Task Willful scale measures attributions of behavior based on willful task avoidance. It ranges from 3 to 18 with higher scores reflecting greater agreement with willful attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 10.14 (0.576) | 10.67 (0.665) | 10.43 (0.576)
  6-Week Follow-up | 9.18 (0.527) | 9.86 (0.608) | 10.89 (0.527)
  12-Week Follow-up | 8.93 (0.576) | 8.57 (0.665) | 10.46 (0.576)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.032, ANOVA; Anova Omnibus F test = 2.723
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .013, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.143; F(2) = 4.595

5. Primary Outcome: Reasons for Children's Behavior - Task Ability Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Task Ability scale measures attributions of behavior based on ability to complete tasks. It ranges from 5 to 30 with higher scores reflecting greater agreement with neurodevelopmental attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 23.29 (0.847) | 22.48 (0.978) | 24.32 (0.847)
  6-Week Follow-up | 22.75 (0.746) | 22.77 (0.862) | 24.57 (0.746)
  12-Week Follow-up | 23.00 (0.922) | 21.57 (1.07) | 23.68 (0.922)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.672, ANOVA; Anova Omnibus F test = 0.588
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .463, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.893; F(2) = .776

6. Primary Outcome: Reasons for Children's Behavior - Disruptive Behavior Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Disruptive Behavior scale measures attributions of behavior based on purposeful disruptive behavior. It ranges from 5 to 30 with higher scores reflecting greater agreement with willful attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 14.96 (1.28) | 17.05 (1.47) | 15.29 (1.28)
  6-Week Follow-up | 12.36 (1.17) | 13.81 (1.35) | 15.50 (1.17)
  12 Week Follow-up | 12.07 (1.25) | 13.24 (1.45) | 14.75 (1.25)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.038, ANOVA; Anova Omnibus F test = 2.612
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .084, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.462; F(2) = 2.544

7. Primary Outcome: Reasons for Children's Behavior - Emotional Support Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Emotional Support scale measures attributions of behavior based on need for emotional support. It ranges from 4 to 24 with higher scores reflecting greater agreement with neurodevelopmental attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 19.50 (0.744) | 20.29 (0.859) | 20.79 (0.744)
  6-Week Follow-up | 20.00 (0.603) | 21.43 (0.697) | 21.43 (0.603)
  12-Week Follow-up | 19.89 (0.636) | 20.91 (0.735) | 21.32 (0.636)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .940, ANOVA; Anova Omnibus F test = 0.196
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .961, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.961; F(2) = .040

8. Primary Outcome: Reasons for Children's Behavior - Dysregulated Behavior Subscale at Baseline, 6-Weeks, and 12-Weeks
Description: The Reasons for Children's Behavior measure assesses parents attributions of behavior. It contains 7 total scales. This Dysregulated Behavior scale measures attributions of behavior based on dysregulated behavior. It ranges from 3 to 18 with higher scores reflecting greater agreement with neurodevelopmental attributions.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 21 | 28
score on a scale
  Baseline | 8.36 (.709) | 9.48 (.819) | 8.964 (.709)
  6-Week Follow-up | 9.43 (.681) | 10.76 (.786) | 10.18 (.681)
  12-Week Follow-up | 8.00 (.717) | 9.38 (.828) | 9.464 (.717)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .671, ANOVA; Anova Omnibus F test = 0.590
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .190, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.523; F(2)=1.696

9. Primary Outcome: Parenting Sense of Competence - Efficacy Sub-scale Baseline, 6-Week, and 12-Week Follow-up
Description: The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The efficacy sub-scale reported here measures how effective parents feel they are and includes 7 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 7 to 42 with higher scores indicating lower feelings of efficacy.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 20 | 28
score on a scale
  Baseline | 26.86 (1.16) | 26.25 (1.37) | 25.32 (1.16)
  6-Week Follow-up | 27.36 (1.15) | 27.15 (1.37) | 25.50 (1.15)
  12-Week Follow-up | 28.39 (1.14) | 29.30 (1.35) | 26.71 (1.14)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .468, ANOVA; Anova Omnibus F test = .896
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .683, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.817; F(2) = .384

10. Primary Outcome: Parenting Sense of Competence - Satisfaction Sub-scale at Baseline, 6-Week, 12-Week Follow-up
Description: The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The satisfaction sub-scale reported here includes 9 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 9 to 54 with higher scores indicating higher satisfaction in the parenting role.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 28 | 20 | 28
score on a scale
  Baseline | 35.36 (1.43) | 32.25 (1.70) | 33.14 (1.43)
  6-Week Follow-up | 36.43 (1.27) | 35.20 (1.50) | 32.68 (1.27)
  12-Week Follow-up | 35.89 (1.39) | 36.15 (1.65) | 32.82 (1.39)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.01, ANOVA; Anova Omnibus F test = 3.42
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .131, Mixed Models Analysis — False discovery rate (FDR) correction for multiple comparisons, p=.480; F(2)=2.081

11. Primary Outcome: Family Needs Questionnaire Baseline to 12-Week Follow-up
Description: The family needs questionnaire measures the degree to which family needs are met. The scale includes 18 items reflecting family needs that are rated on a scale from 0 to 4, with 0 being not applicable to 4 being met a great deal. The total score on this measure is created by summing across all items. Total score ranges from 0-72. Higher scores reflect more needs being met.
Time Frame: baseline to 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 30 | 22 | 29
score on a scale
  Baseline | 40.63 (1.79) | 37.18 (2.09) | 37.93 (1.82)
  12-Week Follow-up | 48.47 (2.07) | 47.00 (2.42) | 42.38 (2.11)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .257, ANOVA; Anova Omnibus F test = 1.384
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .039, Regression, Linear — False discovery rate (FDR) correction for multiple comparisons, p=.055; Cohen's d = 0.49, 95% CI 2-sided [-0.02 to 0.94]

12. Primary Outcome: FASD Knowledge at Baseline and 12-Week Follow-up
Description: The Knowledge and Advocacy questionnaire assesses caregiver knowledge about FASD and advocacy and ranges from 0 to 28. Higher scores reflect greater knowledge.
Time Frame: baseline to 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 30 | 22 | 30
score on a scale
  Baseline | 20.97 (.521) | 21.41 (.609) | 20.73 (.521)
  12-Week Follow-up | 21.30 (.566) | 22.36 (.661) | 20.30 (.566)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .192, ANOVA; Anova Omnibus F test = 1.686
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .039, Regression, Linear — False discovery rate (FDR) correction for multiple comparisons, p=.055; Cohen's d = 0.47, 95% CI 2-sided [0.02 to 0.93]

13. Secondary Outcome: Participant Perception of Self-care Change Over Intervention Period Reported at 12-week Follow-up
Description: Participants are asked at follow-up to rate how much their self-care practices have changed over the last 3 months on a 5-point scale ranging from "A lot less self-care (1)" to "A lot more self-care (5)." A score of 3 equates to no change.
Time Frame: 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
Number analyzed (Participants) | 30 | 22 | 30
score on a scale | 3.10 (1.06) | 3.18 (.795) | 2.90 (.885)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; Mean comparisons of 3 separate groups using ANOVA for 12 week data. Participants with missing data were excluded. All participants were retained in their originally assigned group regardless of app usage; Test type: Superiority; p = .524, ANOVA; Anova Omnibus F test = .651
Statistical Analysis 2: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching) vs Waitlist Comparison Group; The FMF Connect + Coaching and FMF Connect groups were aggregated for analyses. Analyses were intent-to-treat, including all participants assigned to condition. Full information maximum likelihood (FMIL) was used for missing data in MPlus. The dependent variable entered was the measure at the 12-week follow-up to determine treatment effects; Test type: Superiority; p = .048, Regression, Linear — False discovery rate (FDR) correction for multiple comparisons, p=.066; Cohen's d = 0.46, 95% CI 2-sided [0.00 to 0.91]

14. Secondary Outcome: Mean App Quality Score on Mobile App Rating Scale: User Version
Description: The mobile app rating scale includes a measure of users perception of app quality. There are 16 items contributing to this score, each rated on a scale from 1 to 5. Total app quality score is presented as a mean with range of 1 to 5, with higher scores reflecting greater perceived quality of the app.
Time Frame: 12 weeks
Population: Data was analyzed from participants with complete data on the measure from all timepoints. This measure is only applicable to arms that received the app.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching)
Number analyzed (Participants) | 29 | 22
score on a scale | 4.13 (.39) | 4.24 (.32)
Statistical Analysis 1: Comparison: FMF Connect Intervention + Coaching vs FMF Connect Intervention (no Coaching); Test type: Superiority; p = .255, ANOVA; Anova Omnibus F test = 1.32

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events in children with FASD or their caregivers could include aggression or violence towards others, maltreatment, self-harm or suicidality, or the need for inpatient hospitalization. However, these occurrences are unlikely to be a direct consequence of participation in the caregiver intervention or study. These were not systematically assessed but procedures were in place to assess risk and respond appropriately if they arose.
Arm/Group | FMF Connect Intervention + Coaching | FMF Connect Intervention (no Coaching) | Waitlist Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05028517/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05028517/ICF_001.pdf